CLINICAL TRIAL: NCT04874207
Title: Evaluation of Treatment PERSOnalization Based on Its Therapeutic Monitoring in Patients With Metastatic Colorectal Cancer Treated With REgorafenib
Acronym: RePERSO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35RC20_9803_RePERSO
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Patients
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Dose adaptation at the beginning of cycle 2 and cycle 3 after regorafenib dosage at day 15

SUMMARY:
Regorafenib has demonstrated a significant benefit in overall survival in metastatic colorectal cancer (mCRC) patients. However, more than 50% of patients had severe adverse events (grade 3-4), leading to temporary or definitive discontinuation of treatment.

The RePERSO study proposes to adapt the regorafenib dose regimen taking into account firstly the measurement of sum of metabolites M-2 and M-5 and secondly the occurrence of toxicity during treatment. This treatment personalization through therapeutic drug monitoring pharmacological dosing optimization strategy aims at validating the proof of concept of regorafenib therapeutic drug monitoring and at improving the benefit in OS in patients, using the previously defined Csum therapeutic range.

DETAILED DESCRIPTION:
Regorafenib has demonstrated in two multicenter phase III randomized clinical trials a significant benefit in overall survival (OS) in metastatic colorectal cancer (mCRC) patients treated with regorafenib at 160mg/day 3 weeks/4 (3w/4). However, more than 50% of patients had severe adverse events (grade 3-4), leading to temporary or definitive discontinuation of treatment in 2/3 of the patients and a reduction of the dosing in 20% of them. Thus, a part of the therapeutic failures could be explained by an insufficient exposure to regorafenib because of an early toxicity potentially linked to an initial overexposure. The recent randomized phase II ReDOS study has shown that a gradual increase in the dose of regorafenib (from 80 mg to 160 mg/day 3w/4) led to a significantly greater proportion of patients starting a third cycle of regorafenib and showed a trend toward improvement in overall survival of patients when compared to the standard administration schedule (160 mg/day 3 w/4). These results favored the dose-escalation strategy. However, due to the low correlation between dose and concentration, a concentration-controlled study might be of better relevance.

Regorafenib pharmacokinetics is characterized by a hepatic metabolism leading to the production of two main pharmacologically active metabolites (M-2 and M-5) that may induce therapeutic and adverse effects. The production of these metabolites shows a large inter-individual variability. Pharmacokinetic data from phase III studies have suggested the existence of a relationship between exposure to regorafenib and its metabolites and the occurrence of some therapeutic and adverse effects. In an ancillary pharmacokinetic study of the phase II prospective TEXCAN study in which regorafenib was evaluated in its mCRC indication, it was shown a major benefit in OS in patients with an accumulation of M-2 between the first (C1) and the second (C2) cycle of regorafenib (M2 C2/C1). A significant correlation between M-2 C2/C1 ratio and the sum of trough concentrations of regorafenib, M-2 and M-5 measured at D15C1 (C Sum (Rego+M-2+M-5)) was found, which could be a pharmacological marker of efficacy, earlier than the M-2 C2/C1 ratio. The assessment of the relationship between C Sum and in OS according to a Restricted Cubic Spline analysis showed that the benefit is optimal for a concentration between 2.5 mg/L and 5.5 mg/L (median OS of 10.6 months versus 3.3 and 4.0 months in patients with a concentration <2.5 mg/L and ≥5.5 mg/L, respectively). The rate of serious adverse events was also lower in the group in the range [≥2.5; <5.5 mg/L] (0% vs 43% and 20% respectively). This interval seems to allow limiting the severe toxicities that cause treatment discontinuations and/or early progressions that could explain the over-risk of death when the concentrations are outside.

The RePERSO study proposes to adapt the regorafenib dose regimen taking into account firstly the measurement of Csum and secondly the occurrence of toxicity during treatment. This treatment personalization through therapeutic drug monitoring pharmacological dosing optimization strategy aims at validating the proof of concept of regorafenib therapeutic drug monitoring and at improving the benefit in OS in patients, using the previously defined Csum therapeutic range.

ELIGIBILITY:
Inclusion Criteria:

* - Signed and dated informed consent
* Male or female patients ≥ 18 years-old at time of Informed Consent Form (ICF) signature
* Patients must have a histologically proven metastatic colorectal cancer
* Patients who have previously been treated with standard therapy including a fluoropyrimidine, oxaliplatin, irinotecan, an anti-VEGF (bevacizumab or aflibercept) and an anti-EGFR (cetuximab or panitumumab) for patients who had a RAS wild-type tumor
* In mCRC with MSI-H, the patient must have received immunotherapy. For mCRC with BRAF mutation, the patient should have received a BRAF inhibitor if eligible.
* ECOG PS = 0 or 1
* Imaging target greater than one cm must be visible on CT
* Patients must have adequate bone marrow, renal, and hepatic function, as evidenced by the pre-therapeutic check-up performed within 7 days before regorafenib initiation: Normal organ functions as defined below :

  1. Absolute neutrophil count ≥ 1.3 Giga/L
  2. Platelets > 100 Giga/L
  3. Hemoglobin ≥ 9 g/dL
  4. Serum creatinine ≤ 1.5 x ULN (Upper Limit of Normal) or Glomerular filtration rate (GFR) ≥30 ml/min/1.73m2 according to the modified Diet in Renal Disease (MDRD) or CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) abbreviated formula
  5. AST and ALT ≤3 x ULN (≤5.0 × ULN for patients with liver involvement of their cancer)
  6. Total Bilirubin ≤2 X ULN
  7. Alkaline phosphatase ≤3 x ULN (≤5 x ULN in patient with liver involvement of their cancer and/or with bone metastases). If Alkaline phosphatase > 3 ULN (or >5 ULN in patient with liver involvement of their cancer and/or with bone metastases), hepatic isoenzymes 5-nucleotidase or GGT tests must be performed; hepatic isoenzymes 5-nucleotidase must be within the normal range and/or GGT < 3 x ULN
  8. No argument for acute pancreatitis within 3 months before the start of study medication
  9. No proteinuria: Spot urine ≥ 1+ protein will require a 24-hour urine collection that must show total protein excretion <1000 mg/24 hours
* INR/PTT ≤1.5 x ULN
* Patient who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. For patients treated with VKA, close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care
* Women of childbearing potential and male patients must agree to use adequate contraception for the duration of study participation and up to 3 months following completion of therapy
* Women of childbearing potential must have a negative serum β-HCG pregnancy test within 7 days prior randomization
* Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
* Patients affiliated to the Social Security System

Exclusion Criteria:

* - Prior treatment with regorafenib, and with any prior antiangiogenic inhibitor except bevacizumab
* Hypersensitivity to the active substance or to any of the excipients
* Systemic cancer therapy with unfinished washout (in general 3 weeks except for example for capecitabin which has a 1 week washout)
* Concomitant treatment with a cytochrome P450 3A4 (CYP3A4) inducer or inhibitor or UGT1A9 inhibitor
* Patients unable to swallow oral medication
* Digestive obstruction, chronic inflammatory bowel disease or any malabsorption condition
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to inclusion, except for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria])
* Ongoing uncontrolled infection (viral, bacterial or fungal)
* Known history of human immunodeficiency virus (HIV) infection, active hepatitis B or C or chronic hepatitis B or C requiring treatment with antiviral therapy
* Breastfeeding
* Uncontrolled hypertension (systolic blood pressure >140 mmHg or diastolic pressure >90 mmHg despite optimal medical management)
* Arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), within 6 months before the start of study medication
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
* Myocardial infarction less than 6 months before the start of study medication
* Any hemorrhage or bleeding event ≥ Grade 3, NCI-CTCAE v 5.0 within 4 weeks prior to the start of study medication
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days before start of study medication
* Non-healing wound, ulcer or bone fracture
* Unresolved toxicity higher than Grade 1, NCI-CTCAE v 5.0, attributed to any prior therapy/procedure excluding alopecia, anemia, hypothyroidism and oxaliplatin induced neuropathy
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Adults legally protected (judicial protection, guardianship or supervision), person deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Time from inclusion to death | 12 months
  Determine whether "optimal exposure" to regorafenib based on plasma concentration of the drug and its metabolites can improve overall survival in mCRC patients

SECONDARY OUTCOMES:
Ten months survival rate | 10 months
  Percentage of patients alive 10 months after inclusion
Objective response Rate | 12 months
  Objective response Rate (ORR) defined as the rate of patients with complete or partial response
Disease Control Rate | 12 months
  Disease Control Rate (DCR) is defined as the rate of patients with complete response, partial response or stable disease,
Progression-free survival | 12 months
  Progression-free survival (PFS) is defined as the time from inclusion to date of first observed disease progression (radiological or clinical) or death due to any cause, if death occurs before progression is documented. The actual date that the tumor scan was performed will be used for this calculation. PFS for patients without disease progression or death at the time of analysis will be censored at the last date of tumor evaluation.
Severe toxicities | 12 months
  Percentage of patients with significant toxicities (≥ grade 3). Adverse events will be assessed from inclusion to 28 day after the discontinuation of the study drug and classified according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Percentage of optimal exposure | 2 months
  Percentage of patients with "optimal exposure" - i.e. with Csum at day 15 within the range [2.5 - 5.5 mg/L]) - at cycle 1 and cycle 2
Difference in overall survival between patient with different metabolite 2 plasma ratio | 2 months
  Overall survival for the half of patients with a low ratio of plasma concentration of Metabolite 2 Cycle2/Ccyle1 compared to the overall survival for the half of patients with a high ratio of plasma concentration of Metabolite 2 Cycle2/Cycle1
Genetic polymorphism impact | 12 months
  Genetic polymorphisms in gene involved in regorafenib metabolism and plasma concentrations of regorafenib and its metabolites
Body composition | 12 months
  Body composition will be determined on Computerized Tomography scan (CT-scan) imaging done at baseline and for tumor response evaluation during treatment.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Caen, Caen
  - AP-HP Henri Mondor, Créteil
  - Institut Daniel Hollard, Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - CHU Nantes, Nantes
  - AP-HP St Antoine, Paris
  - Centre Eugène Marquis, Rennes
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No